**Project:** Impact Assessment of Triggerise's Tiko Platform (Endline Survey)

Date of Protocol: 25 Feb 2021

**Date of IRB Approval:** 6 March 2021

Consent forms for: (1) Women registered on Tiko (Rafiki) and (2) Tiko Pro

Agents and Service Providers and Shops owners

### Content

| ENGLISH |
|--------------------------------------------|
| Introduction (mention time required) |
| Purpose |
| Sample selection |
| Procedure (mention Time required) |
| Benefits (Service / Compensation / Reward) |
| Risk (Discomfort / Cost / Time) |
| Confidentiality |
| Rights |
| Contact person |
| Consent (Signature / Thumb / Verbal) |

# **Consent Form tiko Platform user young Women**

| <i>Introduction:</i> NAMASTE My name is | | I | am working f | or NEERM | AN, a |
|---|---|---|---|---|---|
| research organization based in Mumba | ii and Delhi. I am her | e to | interview pe | ople on be | ehalf |
| of NEERMAN and Triggerise. | | | | | |

We intend to interview/survey tiko platform user women (mostly age 18-35). The time taken will be approximately 45-50 minutes. I will now give you important details about the survey but please feel free to interject and ask any questions if you may have any.

**Purpose:** In this survey, we intend to collect information on themes of Sexual & Reproductive Health and Maternal health. We would ask you about products and services associated with them (like contraceptives and sanitary pads etc). We also intend to know about your experience with the app you are using —Tiko Explore. This information will be used to help the Triggerise (creator of Tiko Explore) to improve their programs for users like you.

#### Sample selection:

You are one of those users of Tiko Explore who have been chosen by a lottery system to be surveyed and is purely by coincidence and not chosen based on any specifics.

**Procedure:** Once you permit us, we will ask you specific questions on the themes mentioned above. Specifics will include your personal experience and habits of use of products and services associated with the themes. Questions on your experience with Tiko Explore like the ease of use, barriers, or improvements if any will also be asked. Furthermore, we will also ask you questions on your perceptions and outlook, behavior shifts because of the app. Questions around stigma, access, privacy, dignity/respect, willingness to pay, etc will also be asked.

**Benefits of participating in this survey:** There will benefits like a care package of a soap and/or sanitizer costing <Rs 100 or Tiko credit in similar amount to phone-survey respondents. Your inputs and contribution will help the Triggerise, to understand the needs and make any improvements to the platform (Tiko Explore) which might benefit you later. It also greater social good of improving the platform, scaling it up and sustaining it which can benefit others like them.

**Risks of participation:** This study has been approved by a Government-Approved Ethics Committee which will oversee the research to protect study participants as per government guidelines. There are no risks of participating in this survey. But you make have to spare a part of your precious time which may even extend up to 1 hour for this interview. Some of the questions related to contraceptives, pregnancy, family planning can be perceived as too private or invasive. You have the right to refuse answer to such questions. we assure you that all your answers will be kept confidential.

Confidentiality of data and answers: Qualitative interviews will be audio recorded along with notes, quantitative interviews will be conducted using CAPI/CATI apps, and both interviews will collect identifiable information such as name and phone number for survey management purposes only. All the information you share with me is going to be completely confidential. Before giving the data to researchers, we remove all the names, addresses, or any such information that can be linked to you. However, the respondent name, the address, contact information is stored separately. The identification and contact information data will never be given out for any other purpose except for research. Therefore, no one will ever know which person gave what answer. All this is meant to relieve you of any reservations so that that you can give true and organic answers to my questions.

**Respondent's rights:** As a respondent, you have the right not to answer any question you don't want to or you can refuse participation in this survey any time before or during the survey. But, whether or not you choose to participate in this research and whether or not you choose to answer any questions or continue participating in the project, there will be no penalty to you or loss of benefits to which you are otherwise entitled.

**Contact person:** If you have any questions or doubts regarding this survey you can ask me now. If I am unable to answer your questions you can contact Mr. Sagar Kadam, Project Manager of NEERMAN, on 022-24021757 or <a href="mailto:sagar@neerman.org">sagar@neerman.org</a>. If you have any complaints or want to reach higher authority on this you can reach to Karesa Ethics Committee at (+91-80-26667707) <a href="mailto:karesaethics@gmail.com">karesaethics@gmail.com</a>

**Consent:** Your participation in this study is voluntary. Please take your time to make your decision. So, if you want to permit this interview then answer "yes" and please read out the below sentence loudly:

The researcher read to me orally the consent form and explained to me and I agreed to take part in this research.

| (Respondent's Signature) | |
|-----------------------------------------|----------|
| Respondent's Name | Date |
| (Signature of Person Obtaining Consent) | |
| Name of the Person Obtaining Consent | <br>Date |

# Consent Form for Tiko Pro Agents and Service Providers and Shops owners

*Introduction:* NAMASTE. My name is \_\_\_\_\_\_. I am working for NEERMAN, a research organization based in Mumbai. I have come to interview on behalf of NEERMAN and Triggerise.

**Purpose of the survey:** The main aim of our study is to find out the health impact of the Tiko Explore app and its benefits to the participants and actors involved. We interview all the actors involved i.e., users, tiko pro agents, health service providers, shop and service owners demand creators. The questions we ask them will be specific to their role in this ecosystem. The interview/survey will be on themes on Sexual & Reproductive Health, Maternal & Child Health. We also intend to know about your experience with Tiko Explore. This information will be used to help the Triggerise (creator of Tiko Explore) to improve their programs for participants like you.

# (1) Respondent Type: Health Mobilizers (Tiko Pro Agents) and Demand Creators (mass media outlets, peer mobilizers, digital marketers)

Sample selection and Procedure: You are selected for this survey because you are a Tiko Pro Agent who engages with potential users and enroll them onto the platform. There are many eligible agents like you but your selection in this survey has happened through a lottery process and hence only a coincidence. Upon receiving your permission, we will talk to you in detail about your work. You can expect questions like how you engage with the potential users, what training you have got, whether you have been given a phone or tablet, how does it benefit you in your work, how much money were you able to make. We will also talk about your social and economic situation and your experience with Tiko Explore if you have any suggestions and changes to be made.

#### (2) Respondent Type: Product Suppliers(shops, retailers) and Life Style partners (salons, classes)

Sample selection and Procedure: You are selected for this survey because you are one of the service and goods providers to the users who reach you via the Tiko Explore app. We would want to know about your experience with Tiko Explore in how it has affected you and your business and the user experience of the app. You can expect questions like how do you engage with customers and users and the kind of footfall (increase or decrease) you experienced in recent times, to know about the behavior of users who buy goods and services from you among many other questions. Furthermore, we might also ask you questions about the users, their attitudes towards you, the follow-ups, the most common problems they seek your consultation for, etc among many other questions.

#### (3) Respondent Type: Service providers (clinics, pharmacies, hospitals, and healthcare workers)

Sample selection and Procedure: You are selected for this survey because you are one of the several healthcare service providers to the users who reach you via the Tiko Explore app. We would want to know about your experience with Tiko Explore in how it has affected you and your business and the user experience of the app. You can expect questions like how do you engage with customers and users and the kind of footfall (increase or decrease) you experienced in recent times, to know about the behavior of users who buy goods and services from you among many other questions. Furthermore, we might also ask you questions about the users, their attitudes towards you, the goods and services which are popular amongst them among other questions.

**Benefits of participation:** There will not be any tangible benefits (like money, gift voucher, discount voucher) to you personally by participating in this survey. Instead, your inputs and contribution will

help the Triggerise to understand the needs and make any improvements to the platform (Tiko Explore) which might benefit you later.

**Risks of participation:** This study has been approved by a Government-Approved Ethics Committee which will oversee the research to protect study participants as per government guidelines. There are no risks of participating in this survey. But you make have to spare a part of your precious time which may even extend up to 1 hour for this interview. Some of our questions are personal and you may feel hesitant to answer them. Some questions might make you think if the answer to them might affect your business privacy. All your answers are meant and will be used to make the experience better. We assure you that all your answers will be kept confidential.

Confidentiality of data and answers: We also want to inform you that not only is all your information confidential, but you also have some rights as a respondent. The information given to us will be collected in the form of numbers only and will be aggregated to the entire state/village level, but your identity such as name or address will not be given to anyone and will be destroyed. If your interview is audio-recorded with your permission, then the recording is used only to help us finalize the notes and destroyed once the report is written. We may keep this data for the next few years/months for research purposes only. Your data will remain as a number and will be kept secure in a computer with a password.

**Respondent rights:** As a respondent, you have the right not to answer any question you don't want to or you can refuse participation in this survey any time before or during the interview. But, whether or not you choose to participate in this research and whether or not you choose to answer any questions or continue participating in the project, there will be no penalty to you or loss of benefits to which you are otherwise entitled. I can only request you to oblige us by giving your valuable time to this important study.

**Any query:** If you have any questions or doubts regarding this survey you can ask me now. If I am unable to answer your questions you can contact Mr. Sagar Kadam, Project Manager of NEERMAN, on 022-24021757 or <a href="mailto:sagar@neerman.org">sagar@neerman.org</a>. If you have any complaints or want to reach higher authority on this you can reach to Karesa Ethics Committee at (+91-80-26667707) <a href="mailto:karesaethics@gmail.com">karesaethics@gmail.com</a>

Your participation in this study is voluntary. Please take your time to make your decision. So, if you want to permit this interview then answer "yes" and please read out the below sentence loudly:

The researcher read to me orally the consent form and explained to me and I agreed to take part in this research.

| (Respondent's Signature) | |
|-----------------------------------------|------|
| Respondent's Name | Date |
| (Signature of Person Obtaining Consent) | |
| Name of the Person Obtaining Consent | Date |